CLINICAL TRIAL: NCT02025127
Title: A Randomized Controlled Study of Enteral Nutrition in Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Jayshil J. Patel, MD, Principle Investigator, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19966
Record Dates: First submitted 2013-12-17; First posted 2013-12-31 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Septic Shock
Keywords: septic shock; mechanical ventilation; enteral nutrition; trophic feeding
MeSH Terms: conditions — Shock, Septic | interventions — Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trophic feeding (Experimental): Mechanically ventilated patients with septic shock > 18 years old randomized to this group will receive more than 50 but less than 600 kilocalories of enteral nutrition per day while on vasopressors. This will be started within 24 hours of intensive care unit admission.
  Interventions: Other: Enteral nutrition
- No Enteral Nutrition (No Intervention): Mechanically ventilated patients with septic shock randomized to this group will receive no enteral nutrition while on vasopressor support.

INTERVENTIONS:
Other: Enteral nutrition — Enteral nutrition introduced via a feeding tube
  Arms: Trophic feeding

SUMMARY:
There is a paucity of data on the timing and role of enteral nutrition in septic shock.

The primary aim of this study is to conduct a phase III single-center pilot randomized controlled trial comparing early trophic enteral nutrition to 'no enteral nutrition' in mechanically ventilated septic shock patients to determine feasibility.

DETAILED DESCRIPTION:
Septic shock represents the body's dysregulated response to an infection, manifesting as persistent hypotension (mean arterial pressure < 70 mmHg) despite intravenous (IV) fluid resuscitation. Severe sepsis and septic shock are major healthcare problems, affecting millions of people around the world each year In critically ill patients without shock, provision of enteral nutrition within 24-48 hours has shown to preserve intestinal epithelium, maintain brush border enzyme activity, maintenance of barrier function to enhance immune function, and preservation of tight cell junctions to reduce permeability. These benefits of enteral nutrition are postulated to prevent downstream complications of nosocomial infections and the multiple organ dysfunction syndrome (MODS), though direct data addressing this question are lacking.

The primary aim of this study is to conduct a phase III single-center pilot randomized controlled trial comparing early trophic EN to 'no EN' in mechanically ventilated septic shock patients to determine feasibility of achieving >75% consent and compliance rate and <10% contamination rate.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than or equal to 18 years old
* Clinical diagnosis of septic shock
* Mechanically ventilation anticipated for at least 48 hours

Exclusion Criteria:

* Do not resuscitate order
* Not able to obtain consent
* Those not able to be randomized within 18 hours
* Those with small bowel ischemia or obstruction
* Protracted ileus, intractable vomiting, major gastrointestinal bleeding defined as needing 2 or more units of packed red cells, and any bowel surgery within the previous 30 days prior to intensive care unit admission
* Those with a contraindication for placement of a feeding tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-01; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
number of patients consenting to study and remaining compliant with assigned study arm | 46 months
  consent and compliance rate of >75% and contamination rate <10%

SECONDARY OUTCOMES:
Ventilator free days | 30 days
  Number of days alive and off mechanical ventilatory support out of 30
Hospital mortality | 30 days
  number of patients who died during hospitalization
intensive care unit free days | 30 days
  number of days alive and out of the intensive care unit out of 30
change in 48 hour sequential organ failure assessment score, with higher score representing worse outcome | 48 hours
  absolute change in sequential organ failure assessment score (range 0-24 points) from day 0 to 48 hours, with higher scores representing worse outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Jayshil J Patel, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Annane D, Bellissant E, Cavaillon JM. Septic shock. Lancet. 2005 Jan 1-7;365(9453):63-78. doi: 10.1016/S0140-6736(04)17667-8. PMID 15639681
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb S, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including The Pediatric Subgroup. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock, 2012. Intensive Care Med. 2013 Feb;39(2):165-228. doi: 10.1007/s00134-012-2769-8. Epub 2013 Jan 30. PMID 23361625
- [Background] McClave SA, Martindale RG, Vanek VW, McCarthy M, Roberts P, Taylor B, Ochoa JB, Napolitano L, Cresci G; A.S.P.E.N. Board of Directors; American College of Critical Care Medicine; Society of Critical Care Medicine. Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Adult Critically Ill Patient: Society of Critical Care Medicine (SCCM) and American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.). JPEN J Parenter Enteral Nutr. 2009 May-Jun;33(3):277-316. doi: 10.1177/0148607109335234. No abstract available. PMID 19398613
- [Background] Cresci G, Cue J. The patient with circulatory shock: to feed or not to feed? Nutr Clin Pract. 2008 Oct-Nov;23(5):501-9. doi: 10.1177/0884533608323431. PMID 18849555
- [Background] Revelly JP, Tappy L, Berger MM, Gersbach P, Cayeux C, Chiolero R. Early metabolic and splanchnic responses to enteral nutrition in postoperative cardiac surgery patients with circulatory compromise. Intensive Care Med. 2001 Mar;27(3):540-7. doi: 10.1007/s001340100855. PMID 11355123
- [Background] Khalid I, Doshi P, DiGiovine B. Early enteral nutrition and outcomes of critically ill patients treated with vasopressors and mechanical ventilation. Am J Crit Care. 2010 May;19(3):261-8. doi: 10.4037/ajcc2010197. PMID 20436064
- [Background] Bone RC, Balk RA, Cerra FB, Dellinger RP, Fein AM, Knaus WA, Schein RM, Sibbald WJ. Definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. The ACCP/SCCM Consensus Conference Committee. American College of Chest Physicians/Society of Critical Care Medicine. Chest. 1992 Jun;101(6):1644-55. doi: 10.1378/chest.101.6.1644. PMID 1303622